CLINICAL TRIAL: NCT05936567
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging, Efficacy, and Safety Study of Povorcitinib in Participants With Chronic Spontaneous Urticaria
Brief Title: Study Evaluating the Efficacy and Safety of Povorcitinib in Adults With Chronic Spontaneous Urticaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB54707-207; 2022-503062-72-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-06-26; First posted 2023-07-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Urticaria; Chronic Spontaneous Urticaria; Chronic Idiopathic Urticaria; Hives; Angioedema; Pruritis
MeSH Terms: conditions — Urticaria; Chronic Urticaria; Angioedema; Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Povorcitinib Dose A (Experimental): Participants will receive dose A of povorcitinib for a 12 week period, followed by dose A for an additional 24 week period.
  Interventions: Drug: Povorcitinib
- Povorcitinib Dose B (Experimental): Participants will receive dose B of povorcitinib for a 12 week period, followed by dose B for an additional 24 week period.
  Interventions: Drug: Povorcitinib
- Povorcitinib Dose C (Experimental): Participants will receive dose C of povorcitinib for a 12 week period, followed by dose C for an additional 24 week period.
  Interventions: Drug: Povorcitinib
- Placebo followed by Povorcitinib Dose A, B, or C (Experimental): Participants will receive placebo for a 12 week period, followed by randomization to either Dose A, Dose B, or Dose C for an additional 24 week period.
  Interventions: Drug: Povorcitinib; Drug: Placebo

INTERVENTIONS:
Drug: Povorcitinib — oral; tablet
Drug: Placebo — oral; tablet
  Arms: Placebo followed by Povorcitinib Dose A, B, or C

SUMMARY:
This study is being conducted to evaluate the efficacy and safety of povorcitinib in adults with CSU that is inadequately controlled using SOC treatments.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* CSU diagnosis for ≥ 3 months prior to screening.
* CSU refractory to second-generation H1 antihistamines
* Participants must have been on a stable dose of second-generation H1 antihistamine, and must agree to maintain the stable dose of second-generation H1 antihistamine throughout study.
* Willingness and ability to comply with the study Protocol and procedures.
* Further inclusion criteria apply

Exclusion Criteria:

* Treatment with an anti-IgE biologic (eg, omalizumab) within 8 weeks prior to screening.
* Clearly defined underlying etiology for chronic urticarias other than CSU
* Other cutaneous or systemic diseases with chronic itching or with symptoms of urticaria or angioedema.
* Women who are pregnant (or who are considering pregnancy) or breastfeeding.
* Concurrent or history of Thrombocytopenia, coagulopathy, or platelet dysfunction, Venous and arterial thrombosis, deep vein thrombosis, pulmonary embolism, stroke, moderate to severe heart failure (NYHA Class III or IV), cerebrovascular accident, MI, coronary stenting, or CABG surgery, other significant cardiovascular diseases or uncontrolled hypertension
* Recipient of an organ transplant that requires continued immunosuppression.
* Any malignancies or history of malignancies with the exception of adequately treated or excised nonmetastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
* Chronic or recurrent infectious disease.
* Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the urticaria activity score (UAS7) | 12 Weeks
  Defined as the 7-day sum of the individual, daily recorded scores for HSS and ISS, at week 12. UAS scores range from 0-42; with higher scores reflecting greater disease activity.

SECONDARY OUTCOMES:
Proportion of participants who achieve UAS7 ≤ 6 (controlled disease) at Week 12 | 12 Weeks
  Defined as the 7-day sum of the individual, daily recorded scores for HSS and ISS, at week 12. UAS scores range from 0-42; with higher scores reflecting greater disease activity.
Time to first achievement of UAS7 ≤ 6 (controlled disease) during the PC period | 12 Weeks
  Defined as the 7-day sum of the individual, daily recorded scores for HSS and ISS. UAS scores range from 0-42; with higher scores reflecting greater disease activity.
Proportion of participants with UAS7 = 0 at Week 12. | 12 Weeks
  Defined as the 7-day sum of the individual, daily recorded scores for HSS and ISS, at week 12. UAS scores range from 0-42; with higher scores reflecting greater disease activity.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (22):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Cahaba Dermatology, Birmingham, Alabama
  - Foothills Research Center, Scottsdale, Arizona
  - Little Rock Allergy Asthma, Pa Clinical Research Center Lraac, Little Rock, Arkansas
  - Arkansas Research Trials, North Little Rock, Arkansas
  - First Oc Dermatology, Fountain Valley, California
  - Newport Native Md, Newport Beach, California
  - Antelope Valley Clinical Trials Lancaster Office, Palmdale, California
  - Allergy and Asthma Consultants, Pc, Redwood City, California
  - Treasure Valley Medical Research, Boise, Idaho
  - Midwest Allergy Sinus Asthma, Sc, Normal, Illinois
  - Delricht Research, New Orleans, Louisiana
  - David Fivenson, Md, Dermatology, Pllc, Ann Arbor, Michigan
  - Revival Research Institute, Llc Troy, Troy, Michigan
  - The Clinical Research Center Crc, Llc, St Louis, Missouri
  - Optimed Research Ltd, Columbus, Ohio
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, Pc Vpcri, Tulsa, Oklahoma
  - Dermdox Center For Dermatology, Sugarloaf, Pennsylvania
  - Allergy and Asthma Center of Charleston, Charleston, South Carolina
  - Rainey and Finklea Dermatology, San Antonio, Texas
  - Bellingham Asthma, Allergy Immunology Clinic, Bellingham, Washington
- Germany (9):
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Carl Gustav Carus Tu Dresden, Dresden
  - Universitatsklinikum Frankfurt, Frankfurt
  - Mensingderma Research Gmbh, Hamburg
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Universitatsklinikum Leipzig Aor, Leipzig
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Klifos - Klinische Forschung Osnabruck, Osnabrück
  - Universitats-Hautklink Tubingen, Tübingen
- Poland (11):
  - Specderm Poznanska, Bialystok
  - Centrum Medyczne Pratia Katowice I, Katowice
  - Centrum Alergologii Sp Z.O.O, Lublin
  - University Clinical Hospital, Opole
  - Solumed Centrum Medyczne, Poznan
  - Specjalistyczny Nzoz Alergologia Plus, Poznan
  - DC-MED, Swidnica
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych Administracji, Warsaw
  - Etg Warszawa, Warsaw
  - Klinika Ambroziak, Warsaw
  - Melita Medical Sp. Z O. O., Wroclaw

REFERENCES:
- See also: Study Evaluating the Efficacy and Safety of Povorcitinib in Adults With Chronic Spontaneous Urticaria — https://www.incyteclinicaltrials.com/study/?id=INCB54707-207&SearchTerm=INCB54707-207&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=